CLINICAL TRIAL: NCT07239180
Title: Clinical Evaluation of Tunneled Coronally Advance Flap (TCAF) Versus Modified Coronally Advanced Tunnel With Connective Tissue Graft in Management of Single Recession Defects (RT2): A Randomized Clinical Trial
Brief Title: Clinical Evaluation Comparing Tunneled Coronally Advanced Flap and Modified Coronally Advanced Tunnel With Connective Tissue Graft for Managing Single Gum Recession
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khaled Hashem Kamal, Bachelor Degree, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CairoU PhD protocol for Khaled
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Single Recession Defects (RT2)
Keywords: Single Recession defects (RT2); TCAF; MCAT; Clinical performance; Root Coverage; Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Coronally Advanced Tunnel with Connective Tissue Graft (Active Comparator)
  Interventions: Procedure: Modified Coronally Advanced Tunnel with Connective Tissue Graft
- Tunneled Coronally Advance Flap (TCAF) with Connective Tissue Graft (Experimental)
  Interventions: Procedure: Tunneled Coronally Advance Flap with Connective Tissue Graft

INTERVENTIONS:
Procedure: Modified Coronally Advanced Tunnel with Connective Tissue Graft — Modified coronally advanced tunnel with connective tissue graft without vertical releasing incisions
  Arms: Modified Coronally Advanced Tunnel with Connective Tissue Graft
Procedure: Tunneled Coronally Advance Flap with Connective Tissue Graft — Tunneled coronally advance flap with connective tissue graft with one vertical releasing incision
  Arms: Tunneled Coronally Advance Flap (TCAF) with Connective Tissue Graft

SUMMARY:
The technique under investigation aims to provide effective root coverage while offering the advantage of being less invasive.

DETAILED DESCRIPTION:
Limited RCTs have been found in the literature comparing the root coverage capacity of the tunneled coronally advanced flap versus modified coronally advanced tunnel combined with connective tissue graft in single RT2 defects. So, this trial aims to fill this gap of knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Patients with single RT2 gingival recession defect ≥ 2 mm
* Age >18 years old.
* Systemically healthy patients with no contraindications for periodontal surgeries.
* Gingival and plaque index less than 20%.
* No previous surgeries at the defect site.
* Accepts 6 months follow-up period (compliant patients).

Exclusion Criteria:

* RT1 gingival recession.
* Smokers >10 cigarettes a day a contraindicating for any plastic periodontal surgery.
* Poor oral hygiene.
* Active periodontitis patients.
* Patients on medications causing gingival enlargement.
* Pregnancy.
* Teeth mobility ≥ 1 mm.
* Patients using fixed or removable orthodontic appliances.
* Restoration and/or periapical radiolucency at the defect site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-14 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Gingival Recession Depth (GRD) | 6 months
  Measuring gingival recession depth (GRD) using UNC Periodontal probe in millimeter (mm)

SECONDARY OUTCOMES:
The Percentage of Mean Root Coverage (MRC %) | 6 months
  Measuring the percentage of mean root coverage (MRC %) using UNC Periodontal Probe in percentage (%)
Complete Root Coverage (CRC) | 6 months
  Measuring the complete root coverage (CRC) visually (Yes/No)
Root Coverage Esthetic Score (RES) | 6 months
  Measuring the root coverage esthetic score (RES) visually with score (0 "minimum" - 10 "maximum")
The Distance between the contact point and the top of the papilla (DCP) | 6 months
  Measuring the distance between the contact point and the top of the papilla (DCP) using UNC periodontal probe in millimeter (mm)
Gingival Recession Width (RW) | 6 months
  Measuring the gingival recession width (RW) using UNC periodontal probe in Millimeter (mm)
Probing Pocket Depth (PPD) | 6 months
  Measuring the probing pocket depth (PPD) using UNC periodontal probe in Millimeter (mm)
Clinical Attachment Level (CAL) | 6 months
  Measuring the clinical attachment level (CAL) using UNC periodontal probe in Millimeter (mm)
Gingival Index (GI) | 6 months
  Measuring the gingival index (GI) using UNC periodontal probe with score (0 "minimum" - 3 "maximum")
Plaque Index (PI) | 6 months
  Measuring the plaque index (PI) using UNC periodontal probe with score (0 "minimum" - 3 "maximum")
Keratinized Tissue Width (KTW) | 6 months
  Measuring the keratinized tissue width (KTW) using UNC periodontal probe in Millimeter (mm)
Gingival Thickness (GT) | 6 months
  Measuring the gingival thickness (GT) using endodontic file in Millimeter (mm)
Postoperative Patient Satisfaction (Visual Analogue Scale) | 6 months
  Measuring the postoperative patient satisfaction (Visual Analogue Scale) using Patient's questionnaire with score (0 "minimum" -10 "maximum")

IPD SHARING:
Plan to Share IPD: Yes
Limited RCTs have been found in the literature comparing the root coverage capacity of the tunneled coronally advanced flap versus modified coronally advanced tunnel combined with connective tissue graft in single RT2 defects. So, this trial aims to fill this gap of knowledge.

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35175005/